CLINICAL TRIAL: NCT06631768
Title: Gendered Misallocation of Labor: Evidence From Malawian Farmers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nicholas Rahim (Other)
Responsible Party: Sponsor-Investigator, Nicholas Rahim, PhD student in the Department of Global Health and Population, Harvard School of Public Health (HSPH)
Organization: Harvard School of Public Health (HSPH) (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: IRB24-1234
Record Dates: First submitted 2024-10-01; First posted 2024-10-08 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: Maternal and Child Health Outcomes
Keywords: Agriculture; Maternal and child health; Social networks

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment arm with casual labor voucher program (Experimental): Eligible members (pregnant and/or mother of at least one child aged 1 years or younger) of 1AF in the randomly selected treatment districts receive vouchers for a set number of days of free work from casual laborers employed by local 1AF offices. This is in addition to standard 1AF programming.
  Interventions: Other: Casual labor subsidy
- Control arm (No Intervention): Eligible members will only receive standard 1AF programming in randomly selected control districts. They will not receive the labor subsidy during the study period.

INTERVENTIONS:
Other: Casual labor subsidy — Eligible participants will be offered a voucher that can be redeemed for a set number of days of agricultural labor from casual laborers hired by local One Acre Fund offices. Casual laborers receive standard training in line with the trainings currently offered by the organization to participating farmers.
  Arms: Treatment arm with casual labor voucher program

SUMMARY:
The investigators will conduct a cluster randomized controlled trial across districts in Malawi to evaluate the effect of providing free casual labor to pregnant farmers and female farmers on agricultural output, maternal and child health outcomes, child development, and social networks.

DETAILED DESCRIPTION:
This will be a cluster randomized control trial (RCT), where 75 of the districts in which One Acre Fund (1AF) currently operates within in Malawi will be randomly selected for inclusion in this study. Of these 75 districts, 38 will be randomly selected to implement the intervention. The intervention constitutes a voucher offered to all female famers who are currently enrolled in the 1AF program who are pregnant and/or have a child ages 1 years and below that entitles the recipient to a set number of days of labor from casual workers employed by local 1AF offices. The remaining 37 districts will serve as the control group.

Data will be collected at baseline during the planting season and endline at the conclusion of the harvest season. Data collected will pertain to agricultural output, individual and household demographics, obstetric history and outcomes, mental health, maternal health, child health and development, and social networks.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant at time of One Acre Fund program rollout
* Mother to at least one child aged below 1 years of age

Exclusion Criteria:

-None

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 989 (Actual)
Dates: Start 2025-08-16 (Actual); Primary Completion 2025-09-07 (Actual); Study Completion 2025-09-07 (Actual)

PRIMARY OUTCOMES:
Agricultural Output | Assessed after harvest season (6 - 8 months after intervention initiation)
  A continuous measure of the value of the participant's agricultural yield, measured in Malawian Kwacha
Labor inputs | Assessed after harvest season (6 - 8 months after intervention initiation)
  A pair of recall questions repeated for each household member aged 10 years or older (including the respondent) that ask about the average number of days a week and the average number of hours per day the individual works on the respondent's farm, both measured continuously.
Antenatal care seeking | Assessed after harvest season (6 - 8 months after intervention initiation)
  A continuous variable of number of antenatal care visits for those pregnancies that overlap with the index agricultural season
Care seeking for child health | Assessed after harvest season (6 - 8 months after intervention initiation)
  Two continuous variables measuring number of routine postnatal care and sick child visits
Reach of social networks | Assessed after harvest season (6 - 8 months after intervention initiation)
  A social networks module that collects data on the extent and characteristics of the participant's social networks. Measured by the number of people reported in the participant's network, with a higher number indicating a larger network.
Postnatal care seeking | Assessed after harvest season (6 - 8 months after intervention initiation)
  A continuous variable of number of postnatal care visits for those pregnancies that overlap with the index agricultural season

SECONDARY OUTCOMES:
Maternal consumption short term recall: number of meals | Assessed after harvest season (6 - 8 months after intervention initiation)
  Two questions regarding the number of meals consumed the day before and the number of meals consumed two days before
Maternal consumption medium term recall: protein intake | Assessed after harvest season (6 - 8 months after intervention initiation)
  Four questions regarding the number of times the participant consumed fish, meat, eggs, and usipa.
Maternal mental health | Assessed after harvest season (6 - 8 months after intervention initiation)
  Patient Health Questionnaire-2 (PHQ-2): a 2-item Likert scale questionnaire for assessing depressive symptoms. Score can range between 0 and 6, with higher scores indicating more severe depressive symptoms.
Child birth weight | Assessed after harvest season (6 - 8 months after intervention initiation)
  A continuous variable measured in grams of the reported birthweight of each child born during most delivery
Barriers to perinatal care | Assessed after harvest season (6 - 8 months after intervention initiation)
  A set of four Likert style questions asking to respondents to how much they agree with the following statements as reasons to not visit a health facility for ANC and/or PNC: "The health facility is too far away," "I have to work on my farm," "I am too unwell/sick," "and "I do not think the quality of care is worth it"
Maternal hunger | Assessed after harvest season (6 - 8 months after intervention initiation)
  Question about how often the respondent went to bed hungry in the past month: "Never," "A few times," "Nearly every other night," and "Most nights"
Child consumption | Assessed after harvest season (6 - 8 months after intervention initiation)
  A set of four questions concerning the frequency of breastfeeding; meat, egg, or fish; fruits or vegetables; and porridge, bread, rice, pap, or pasta consumption in the past month for the youngest child.
Willingness to hire causal labor | Assessed after harvest season (6 - 8 months after intervention initiation)
  Likert scale question on how likely the participant is to hire a casual worker during the upcoming agricultural season

CONTACTS AND LOCATIONS:
Overall Officials: Gabriella Fleischman, Principal Investigator — Harvard Kennedy School; Nicholas Rahim, Principal Investigator — Harvard School of Public Health (HSPH)
Locations (1):
- One Acre Fund, Zomba, Zomba, Malawi

IPD SHARING:
Plan to Share IPD: Yes
After manuscript publication, fully de-identified data may be shared with researchers upon request.